CLINICAL TRIAL: NCT06819787
Title: Patient-Reported Outcomes of Contraceptive Services Rendered by Community Pharmacists Using the Pharmacist Resource to Implement Services as Modules Platform: The PRISM-CS Study
Brief Title: Patient Experiences With Contraceptive Care Provided by Community Pharmacists Using the Pharmacist Resource to Implement Services as Modules Platform
Acronym: PRISM-CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OvaryIt, LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2R44HD110346-02A1 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Contraception
Keywords: Contraception; Pregnancy Prevention; Digital Health; Pharmacist; Community Pharmacy Services; Patient-reported Outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacist-Rendered Contraceptive Services (Experimental): Participants in this single-arm study are women seeking contraceptive services to prevent pregnancy in a community pharmacy setting. Pharmacists will deliver these services using an Electronic Health Record system that assists in evaluating each patient's eligibility based on the US Medical Eligibility Criteria (USMEC) guidelines. Pharmacists will be instructed to provide patient-centered contraceptive care. They retain full discretion to decide whether to issue a prescription, and if so, to select the most appropriate FDA-approved contraceptive option based on their clinical judgment.
  Interventions: Other: Electronic Heath Record Platform to Support Pharmacists in Delivering Contraceptive Services

INTERVENTIONS:
Other: Electronic Heath Record Platform to Support Pharmacists in Delivering Contraceptive Services — An electronic health record (EHR) platform specifically designed to support community pharmacists in delivering contraceptive services. The platform streamlines clinical workflows, provides clinical decision support, and promotes adherence to the US Medical Eligibility Criteria (USMEC) guidelines and state regulatory requirements.

SUMMARY:
Hormonal contraceptives are medications that require a prescription, traditionally from a physician or advanced practice provider. Over the past decade, pharmacists have gained the authority to prescribe contraceptives in many states, allowing patients to access these medications directly in pharmacies without first seeing another healthcare provider. The Pharmacist Resource to Implement Services as Modules (PRISM) is an Electronic Health Record platform designed to streamline workflows and provide clinical decision support, making it easier and safer to deliver clinical services in community pharmacies. This pilot study will evaluate patient-reported outcomes for women receiving contraceptive services from pharmacists using the PRISM platform at five community pharmacies across the United States over a 12-week period. The study will assess the quality of care, contraception continuation and failure rates, side effect rates, preventative healthcare utilization, and overall patient experience with pharmacy contraceptive services.

ELIGIBILITY:
Inclusion Criteria:

• Women presenting for hormonal contraceptives

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Unable to become pregnant
* Not English speaking
* Suspected coercion
* Unable to consent

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2025-07-12 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Person-Centered Contraceptive Counseling (PCCC) Measure | Within 7 days post-intervention
  The percentage of patients who report that the pharmacist provided overall patient-centered care, as defined by achieving the highest rating on all four items of the PCCC survey.

SECONDARY OUTCOMES:
Three-month Contraceptive Continuation Rate | Within 97 days post-intervention
  The percentage of patients who report continuous use of their selected contraceptive method three months after the pharmacist encounter. Continuous use is defined as using the method at the time of the survey with no gaps in use of one month or longer.

OTHER OUTCOMES:
Contraceptive Failure Rate | Within 97 days post-intervention
  The percentage of patients who have experienced unintended pregnancy while using the contraceptive method prescribed during the encounter.
Contraceptive Side Effect Rate | Within 97 days post-intervention
  The percentage of patients who report one or more side effects from the contraceptive method prescribed during the encounter.
Patient Contraceptive Satisfaction | Within 97 days post-intervention
  7-point Likert scale rating of patient satisfaction with the contraceptive method prescribed during the encounter.
Patient Perception, Attitudes, and Satisfaction Regarding Pharmacist Contraceptive Services | Within 97 days post-intervention
  A series of Likert scale, Yes/No, and open-ended questions to discover patient perceptions, attitudes, and satisfaction regarding pharmacist contraceptive services.
Preventative Health Services Utilization | Within 97 post-intervention
  A series of Yes/No and multiple-choice questions to discover patient utilization of preventative health services including primary care and medical screening exams.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Calabasas Pharmacy, Calabasas, California
  - Desert Pharmacy, El Centro, California
  - Local Health Pharmacy, Chicago, Illinois
  - Wolves Den Pharmacy, Stanford, Montana
  - Gaston Family Pharmacy, Gaston, South Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT06819787/ICF_000.pdf